CLINICAL TRIAL: NCT03375346
Title: Effects of Whole-body Vibration Exercise on Brain Activity and Physical Function in Hemiplegia Stroke Patients
Brief Title: Effects of Whole-body Vibration Exercise on Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-07-092
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Stroke; Hemiplegia
Keywords: Whole body vibration exercise
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Eligible patients were randomly assigned to one of the two groups in a 1:1 ratio using an odd or even random numbers table. Whole body vibration group performed a single session of whole body vibration exercise via a vibrating platform (Galileo® Advanced Plus, Novotec Medical, Pforzheim, Germany) with a magnitude of 20 Hz and an amplitude of 4 mm. The control group performed the same session without vibration.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration group (Experimental): Whole body vibration group performed a single session of whole body vibration exercise via a vibrating platform (Galileo® Advanced Plus, Novotec Medical, Pforzheim, Germany) with a magnitude of 20 Hz and an amplitude of 4 mm.
  Interventions: Device: Whole body vibration; Other: Exercise
- Exercise only group (Active Comparator): The control group performed the same session without vibration.
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Whole body vibration — whole body vibration exercise is a stimulus that uses vibrations generated on a machine with oscillatory movement determined by the amplitude and frequency of the vibration.
  Arms: Whole body vibration group
Other: Exercise — maintain a half-squat position (knee joint angle at 160 degrees) on the tilt table with an incline of 60 degrees

SUMMARY:
The purpose of this study is to investigate the effect of the whole body vibration exercise on cortical activity and gait function in patients with chronic stroke.

DETAILED DESCRIPTION:
Whole body vibration exercise can provide proper somatosensory stimulation and improve muscle strength and postural control in stroke patients. However, there has not yet been a report on the cortical activity changes induced by whole body vibration exercise.

Patients will be randomly assigned to one of the two groups. One group will go through whole body vibration with exercise and the other will only perform exercise. The primary outcome measurement of this study was cerebral cortex activity based on changes in oxygenated hemoglobin concentration using functional near-infrared spectroscopy. Behavioral assessments were performed before and after the intervention session using the 10-meter walk test, timed up and go test, Fugl-Meyer Assessment, and Tinetti Performance Oriented Mobility Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke with hemiplegia
* 3 months after stroke onset
* Able to walk at least 10 meters without assistive devices

Exclusion Criteria:

* Subjects under 18 years and above 80 years old,
* Unable to perform a half squat on a vibrator (eg. visual field defects, fracture, and severe muscle paralysis)
* Musculoskeletal disorders
* Risk of falling due to dizziness
* Pregnant women

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Cerebral cortex activity | check before, during and directly after intervention(for approximately 14 minutes)
  cerebral cortex activity was measured based on changes in oxygenated hemoglobin concentration using fNIRS

SECONDARY OUTCOMES:
10 meter walk test | before and after intervention(Approximately 14 minutes)
  performance measure used to assess walking speed in metres per second over a short distance. It can be Blender3D NormalWalkCycle.gifemployed to determine functional mobility, gait, and vestibular function.
Timed up and go test | before and after intervention(Approximately 14 minutes)
  test for gait speed and gait balance
Fugl-Meyer Assessment | before and after intervention(Approximately 14 minutes)
  a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Tinetti Performance Oriented Mobility Assessment | before and after intervention(Approximately 14 minutes)
  Task-oriented outcome measure that assesses gait and balance ability; is composed of a 9-item gait portion (POMA-G) and 7-item balance portion (POMA-B)

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee A, Kim H, Kim J, Choi DS, Jung JH, Lee J, Kim YH. Modulating Effects of Whole-body Vibration on Cortical Activity and Gait Function in Chronic Stroke Patients. Brain Neurorehabil. 2020 Mar 26;13(2):e12. doi: 10.12786/bn.2020.13.e12. eCollection 2020 Jul. PMID 36744184